CLINICAL TRIAL: NCT05164354
Title: The Effect of Cancer Therapy and Music Concert Applied to Children on Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ayse Arıcıoglu Sulun, Dr. Research Asistant, Inonu University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/165
Record Dates: First submitted 2021-11-19; First posted 2021-12-20 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Pediatric Cancer; Sleep
Keywords: Pediatric cancer; sleep; aromatherapy; music concert
MeSH Terms: conditions — Neoplasms | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: NAfter the pre-test is applied to the experimental group, music therapy and aromatherapy will be given to the experimental groups by the researcher.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy (Experimental): Aromatherapy will be done in the form of a 20-minute application period for three days.
  Interventions: Other: Aromatherapy
- music concert (Experimental): "Music concert" will be performed in the form of a 20 minute daily practice period for three days.
  Interventions: Other: music concert

INTERVENTIONS:
Other: Aromatherapy — Aromatherapy: It will be applied to each child three times, three days in a row. Each application will be 20 minutes. The application time will be decided together with the patient. At the end of the three-day practice.
  Arms: Aromatherapy
Other: music concert — Music Concert: In this study, a music (lullaby, classical music) to be preferred by the patient or family Children are played for 20 minutes once a day. (morning or afternoon) for three days to help the child sleep. The volume of the music being played will be preserved. Aromatherapy: To be applied each child three times for three consecutive days. Each one The application will take 20 minutes. It will be time to implement The decision is made with the patient. Finally The patient's sleep quality will increase in three days of application. measured by actigraphy.
  Arms: music concert

SUMMARY:
The actigraph device continuously records the occurrence of limb movements and then collects the number of movements in a given time interval. Compared to polysomnography Actigraphy is a reliable and valid method for monitoring sleep in infants.

DETAILED DESCRIPTION:
Cancer is a disease characterized by rapid proliferation and uncontrollable growth of abnormal cells . According to the tumor statistics data of the Turkish Pediatric Oncology Group (TPOG), the incidence of cancer in children aged 10-14 in Turkey is 22.80 per million (n= 2756), while this rate is 7.35 per million in children aged 15-19 years (n= 2756). 886). Despite the high incidence of cancer, it has started to be seen as a life-threatening chronic disease rather than a terminal disease with the treatment methods developed in the field of pediatric oncology However, early initiation of treatment, effective treatment use, and high treatment success have made increasing the quality of life and psychosocial approach even more important. However, both cancer diagnosis and treatment reduce the child's quality of life and cause many psychosocial and physical problems.

Sleep plays a role in many important functions such as growth and development, tissue regeneration, energy conservation, and strengthening of the immune system in childhood.

Inadequate sleep quality and sleep disorders are frequently observed in children diagnosed with cancer . Sleep problems are seen in approximately half of children with cancer. Difficulty falling asleep, waking up suddenly during sleep, difficulty waking up, and excessive daytime sleepiness are symptoms that indicate inadequate sleep quality in children with cancer .

Sleep problems begin with the diagnosis of children with cancer, and the amount and quality of sleep of the child is negatively affected due to reasons such as unfamiliar environment, deterioration of sleep habits, and staying away from their own bed at the first admission to the clinic. In addition, symptoms such as side effects related to the treatment initiated, disruption of sleep routine due to treatment, and pain due to illness cause sleep problems . These sleep problems make it difficult for children to comply with treatment and reduce their quality of life.

Alternative pharmacological and non-pharmacological methods can be used in the management of cancer-related sleep disorders . Aromatherapy and listening to music are among the recommended non-pharmacological methods .

Arometherapy is a therapy method that is used frequently all over the world and that explores the use of essential oils to treat and protect the health of individuals .

Music concert is one of the methods aimed at improving the health and well-being of individuals. Although it has a positive effect on children physically, psychologically, socially and emotionally, it is an economical and side-effect-free method. No studies have been found in the literature evaluating the sleep status of children with cancer with music therapy.

There are studies in which aromatherapy and music therapy are applied in children with cancer.

Although there are studies reporting that aromatherapy and music therapy are effective in relieving the symptoms of children with cancer. In this direction, there is a need for studies that compare these methods with each other and have a high level of evidence, as well as the effectiveness of aromatherapy and music therapy in children with cancer.

ELIGIBILITY:
Inclusion Criteria:

- Being oriented, open to communication and cooperation

Exclusion Criteria:

- Not in the induction phase of cancer treatment

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Actigraphy device | three days
  The actigraph device continuously records the occurrence of limb movements and then collects the number of movements in a given time interval. Compared to polysomnography Actigraphy is a reliable and valid method for monitoring sleep in infants.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Battalgazi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kutluk T YA. Turkish National Pediatric Cancer Registry 2002-2008. 41st Congress of International Society for Pediatric Oncology. Sao Paulo, Brazil. In: On behalf of Turkish Pediatric Oncology Group and Turkish Pediatric Hematology Society Turkish National Pediatric Cancer Registry 2002-2008 41st Congress of International Society for Pediatric Oncology Sao Paulo, Brazil. 2009. p. 851.
- [Background] Kudubeş AA, Bektas M, Bektas İ, Selekoglu Y, Sal Altan S, Ayar D. The effect of symptom frequency on the fatigue and sleep quality of adolescent cancer patients. Child Heal Care. 2017;46(4):421-38.
- [Background] Walter LM, Nixon GM, Davey MJ, Downie PA, Horne RS. Sleep and fatigue in pediatric oncology: A review of the literature. Sleep Med Rev. 2015 Dec;24:71-82. doi: 10.1016/j.smrv.2015.01.001. Epub 2015 Jan 13. PMID 25679070
- [Background] Kaleyias J, Manley P, Kothare SV. Sleep disorders in children with cancer. Semin Pediatr Neurol. 2012 Mar;19(1):25-34. doi: 10.1016/j.spen.2012.02.013. PMID 22641073
- [Background] Graef DM, Crabtree VM, Srivastava DK, Li C, Pritchard M, Hinds PS, Mandrell B. Sleep and mood during hospitalization for high-dose chemotherapy and hematopoietic rescue in pediatric medulloblastoma. Psychooncology. 2018 Jul;27(7):1847-1853. doi: 10.1002/pon.4737. Epub 2018 May 16. PMID 29663636
- [Background] Kushner BH, LaQuaglia MP, Wollner N, Meyers PA, Lindsley KL, Ghavimi F, Merchant TE, Boulad F, Cheung NK, Bonilla MA, Crouch G, Kelleher JF Jr, Steinherz PG, Gerald WL. Desmoplastic small round-cell tumor: prolonged progression-free survival with aggressive multimodality therapy. J Clin Oncol. 1996 May;14(5):1526-31. doi: 10.1200/JCO.1996.14.5.1526. PMID 8622067
- [Background] Allen JM, Graef DM, Ehrentraut JH, Tynes BL, Crabtree VM. Sleep and Pain in Pediatric Illness: A Conceptual Review. CNS Neurosci Ther. 2016 Nov;22(11):880-893. doi: 10.1111/cns.12583. Epub 2016 Jul 15. PMID 27421251
- [Result] American Cancer Society. Cancer Facts & Figures 2016. Cancer Facts Fig 2016. 2016;1-9.